CLINICAL TRIAL: NCT07186309
Title: A Prospective Validation of the Enlighten Device in Predicting Postpartum Depression Using At-Home Sample Collection in Both Blood and Saliva
Brief Title: A Study of a Test for Postpartum Depression at Home
Acronym: BRAVE
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Mayo Clinic (Other); Dionysus Health (Unknown)
Responsible Party: Principal Investigator, Jennifer L. Payne, Principal Investigator, University of Virginia
Other Study IDs: 20252779; HT94252510260 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Depression (PPD); Pregnancy
Keywords: Pregnancy; Postpartum Depression; Predictive Test; Blood Test; Third Trimester; Behavioral Symptoms; Mood Disorders; Mental Disorders; Puerperal Disorders; Pregnancy Complications; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Depression, Postpartum; Depression; Depressive Disorder
MeSH Terms: conditions — Depression, Postpartum; Behavioral Symptoms; Mood Disorders; Mental Disorders; Puerperal Disorders; Pregnancy Complications; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Depression; Depressive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Saliva Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Diagnostic Test: Enlighten — The primary analysis will examine the performance of the Enlighten Device by evaluating biomarker status results ("elevated risk" or "low risk") at the third trimester against depression symptoms outcome data collected by the 3 months postpartum time point.

SUMMARY:
The study will seek to prospectively validate the Enlighten Device for prediction of PPD by examining true/false positive and negative rates of the test using PPD outcomes collected through 3 months postpartum; compare the accuracy of biomarkers and algorithm in determining risk for PPD in blood compared to saliva; determine the utility of a week 6 sample collection in identifying women who are currently experiencing PPD thus bringing them to clinical attention.

Our population will consist of pregnant women aged 18 and older up to 33 weeks of gestation. This research involves two groups of potentially vulnerable subjects: pregnant women and their infants. Because this is a study of postpartum depression (PPD), inclusion of these two vulnerable subjects is required. The study will enroll 1000 pregnant non-adolescent women of childbearing age who meet eligibility criteria.

This project will address the following Aims:

Specific Aim 1: Prospective collection of true/false positive and negative PPD outcomes through 3 months postpartum.

Primary Hypothesis H1a: 80% or greater of pregnant women who develop postpartum depression (PPD) by 3 months after delivery will be determined to be Biomarker Positive by the Enlighten Test in T3.

Primary Hypothesis H1b: 10% or fewer of pregnant women who are determined to be Biomarker Negative by the Enlighten Test in T3 will develop PPD by 3 months after delivery.

Exploratory Aim 1: Investigation of clinical factors that may be associated with false positive and false negative rates, such as: medication use, stressful life events, & sociocultural context.

Specific Aim 2: Comparison of prospective biomarker calls made in blood samples compared to saliva samples using the Enlighten Test.

Primary Hypothesis H2: Biomarker calls made using blood versus saliva samples will demonstrate a high concordance rate of 75% or higher.

Exploratory Aim 2: In individuals who develop PPD by 3 months postpartum, conduct an epigenome-wide study (EWAS) in saliva to identify saliva-specific epigenetic biomarkers to improve the algorithm's ability to predict PPD using saliva in the third trimester and Week 6 samples.

Specific Aim 3: Determination of the utility of the Enlighten Test in identifying women currently experiencing PPD at W6 postpartum.

Primary Hypothesis H3: 80% of women who meet criteria for PPD at W6 will be Biomarker Positive.

Participants will be screened during the second or third trimester and enrolled during the third trimester, before week 30 weeks of gestation. Participants may self- identify through study advertisements in participating clinics, social media outlets, and community outreach efforts. Enrolled participants will undergo blood collection during their 3rd trimester completed by mobile phlebotomists in-person through ExamOne (~27-30 weeks, a standard pregnancy-related blood collection timepoint) for completion of the Enlighten Device test, the blood-based epigenetic biomarker test. Participants will then be interviewed at 2 weeks, 6 weeks, and 3 months postpartum for the development of depression symptoms. They'll also complete a multitude of other outcome measures at each of these visits.

ELIGIBILITY:
Inclusion Criteria:

* subject must be pregnant (singleton pregnancy)
* <30 weeks' gestation, age 18 or above
* able to provide written consent in English

Exclusion Criteria:

* The study team and/or PI may exclude anyone deemed unsafe to participate in the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 1,000 pregnant women aged 18 and older up to 33 weeks of gestation
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with True/False Positive and Negative PPD Outcomes as Assessed by the Enlighten Device | 6 months postpartum
  PPD diagnosis will be confirmed by clinical evaluation using the Structured Clinical Interview for the DSM-5 Research Version (SCID-5-RV) and Edinburgh Postnatal Depression Scale (EPDS), at the time of enrollment and subsequent study visits. True positive/negative and false positive/negative classifications will be based on the Enlighten Device's biomarker threshold values in T3 (third trimester). Data will be aggregated as percentages and compared to clinical PPD diagnoses.
  Primary Hypothesis H1b: 10% or fewer of pregnant women who are determined to be Biomarker Negative by the Enlighten Device in T3 will develop PPD by 3 months after delivery.
  Exploratory Aim 1: Investigation of clinical factors that may be associated with false positive and false negative rates, such as: medication use, stressful life events, and sociocultural context.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share de-identified data with other researchers. Data shared will include demographic information, clinical data which will include SCID diagnosis, mental health surveys like EPDS, PASS, etc., sample analyses data.
Supporting Information: Study Protocol